CLINICAL TRIAL: NCT02684643
Title: Study of Individualized Therapy on Hyperphosphatemia in Maintenance Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Chen Jing, Chief Physician of Division of Nephrology, Professor, Associate Director of Division of Nephrology and Director of Dialysis Centre, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2015-271
Record Dates: First submitted 2016-01-28; First posted 2016-02-18 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Hyperphosphatemia; End-stage Renal Disease
Keywords: individualised therapy; hyperphosphatemia; hemodialysis; clinical trials; restricted phosphate diet; phosphate binders
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- enhanced individualised therapy (Experimental): Patients' dialysis dosage, medication as well as dietary plan will be modified.
  Interventions: Other: enhanced individualised therapy
- non-enhanced individualised therapy (Experimental): Patients' medication as well as dietary plan will be modified without alteration of dialysis dosage.
  Interventions: Other: non-enhanced individualised therapy
- regular intervention (Experimental): Phosphate binders and calcitriol will be prescribed and adjusted without altering patients' diet habit.
  Interventions: Other: regular intervention

INTERVENTIONS:
Other: enhanced individualised therapy — additional dialysis dosage, modification of medication and prescribed dietary plan
  Arms: enhanced individualised therapy
Other: non-enhanced individualised therapy — modified medication, prescribed dietary plan and regular three times/week dialysis dosage
  Arms: non-enhanced individualised therapy
Other: regular intervention — Phosphate binders and calcitriol would be prescribed according to the guidelines. Phosphate binders included in the study are calcium acetate, calcium carbonate or sevelamer. Dosage is based on patients serum phosphate and calcium level. Calcitriol prescribed in the study is Rocaltrol and the dosage is based on PTH, serum phosphate and calcium level. Patients' diet habit will not be altered.
  Arms: regular intervention

SUMMARY:
This study is designed to study and compare the efficacy and cost-effectiveness of individualized phosphate-lowering therapy in comparison with regular guideline-recommended therapy.

DETAILED DESCRIPTION:
Hyperphosphatemia in hemodialysis patients has been one of the most difficult conundrums for nephrologist for the past two decades. Elevated phosphate contributes to secondary hyperparathyroidism, elevated FGF23 levels, and vascular calcification, which in turn predispose to mortality in this population. Current guidelines recommend limiting dietary phosphate intake, strengthening dialysis and using phosphate binders as three therapies for treatment of hyperphosphatemia. Yet exact clinical implication remains ambiguous: how intense restricted phosphate intake should be and how dosage of phosphate binders and dialysis should be adjusted accordingly. Thus, treatments of hyperphosphatemia have not been effective enough, but appear to be refractory. In the current study, the investigators designed individualized phosphate-lowering therapy based on each patient's phosphate-clearing ability, in order to observe and compare the efficacy and cost-effectiveness of the individualized therapy and the regular guideline-recommended therapy.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70 years' old
* dialysis vintage more than 3 months on maintenance hemodialysis patients
* using internal arteriovenous fistula
* S[P] > 1.45 mmol/l, PTH (parathyroid hormone, PTH) < 900 ng/ml
* no residual renal function (RRF)
* stable dietary habit
* clear consciousness and capable of communication
* willingness to give written consent and comply with the study protocol

Exclusion Criteria:

* severe infection, anemia (Hb < 60 g/L), hypoproteinemia (Alb < 30 g/L)
* pregnancy, lactating women
* history of severe coexisting diseases such as, but not limited to, chronic liver disease, myocardial infection, cerebrovascular accident, malignant hypertension
* history of malignancy
* participation in other dietary, drug-related, or any other clinical trials within 1 month
* history of complications related to elevated S[P] such as, but not limited to primary hypoparathyroidism, type II vitamin D dependent rickets
* history of non-compliance
* intolerance to the individualized therapy
* in use of calcitonin and diphosphonate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2016-01; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Serum phosphate level at the end of the trial | 6 weeks

SECONDARY OUTCOMES:
Serum calcium | 6 weeks
parathyroid hormone | 6 weeks
  serum iPTH level
cost of the therapy | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086